CLINICAL TRIAL: NCT06028386
Title: A Prospective Pilot Study Evaluating Wound Closure With the Application of AC5® Advanced Wound System in the Treatment of Diabetic Foot Ulcers
Brief Title: Use of AC5® Advanced Wound System in the Treatment of Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arch Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-1003
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Non-healing Wound; Diabetic Foot Ulcer
Keywords: DFU; self-assembling peptide; chronic wounds; Synthetic matrix
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1-AC5® Advanced Wound System (Active Comparator): The intervention in this arm is the application of a synthetic self assembling peptide matrix (AC5) to UT Grade 1A diabetic foot ulcers
  Interventions: Device: AC5® Advanced Wound System
- Arm2- Fibracol Plus Collagen dressing (Placebo Comparator): The intervention in this arm is the application of collagen dressings to UT Grade 1A diabetic foot ulcers
  Interventions: Device: Fibracol Plus Collagen Dressing

INTERVENTIONS:
Device: AC5® Advanced Wound System — This group will receive AC5® Advanced Wound system, a synthetic self-assembling peptide matrix to the wound and covered with non-adherent dressing followed with appropriate outer dressing to maintain moisture balance. AC5 is applied weekly and outer dressing will be redressed as necessary.
  Arms: Arm 1-AC5® Advanced Wound System
Device: Fibracol Plus Collagen Dressing — This group will receive Fibracol Plus collagen dressing to the wound and covered with appropriate out dressing. Treatment will be done 3x a week.
  Arms: Arm2- Fibracol Plus Collagen dressing

SUMMARY:
The purpose of this clinical evaluation is to collect and compare outcomes data from patients with UT 1A diabetic foot ulcers treated with 510K FDA cleared, commercially available self-assembling peptide, AC5®Advanced Wound System, as compared to an advanced standard of care. Patient outcomes will be compared at the end of the study.

DETAILED DESCRIPTION:
This study is a prospective, multi-center randomized controlled study designed to collect patient outcomes data for the treatment of diabetic foot ulcers. (DFU) All subjects will receive standard of care procedures (SOC) such as wound cleaning, appropriate sharp debridement, and appropriate offloading of the DFU (e.g., offloading Camboot or post op shoe with offloading/wound care insole).

Subjects will be randomized and receive treatments to either of the following arms:

Arm 1 - Subject will receive SOC that will include AC5® Advanced Wound System as an active synthetic cellular tissue product, covered with a non-adherent dressing plus an appropriate outer dressing to maintain moisture balance, then wrapped with stretch gauze and self-adherent wrap. AC5 will be applied weekly and outer dressings will be redressed, if necessary, using the allowed secondary dressings.

Arm 2 - Subject will receive SOC that will include Fibracol Plus collagen dressing as an active dressing. This will be followed with an appropriate outer dressing to maintain moisture balance, then wrapped with stretch gauze and self-adherent wrap as needed. Fibracol Plus will be applied 3 x a week and any outer dressings will be redressed, if necessary, using the allowed dressings.

The study involves two phases: Screening and Treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 or older.
2. Subject is willing to sign informed consent and participate in all procedures with follow up evaluations as necessary to complete the study.
3. Study ulcer is diabetic in origin, located on the foot or below the malleolus with ulcer extending through the dermis but not into tendon, muscle or bone (UT Grade 1A).
4. Study ulcer size is a minimum of 2 cm2 and maximum 25 cm2 after the run-in period.
5. Study ulcer has been present for a minimum of 4 weeks before enrollment and less than 1 year old, with documented failure of prior treatment to heal the wound.
6. Study ulcer has been offloaded for at least 14 days prior to randomization.
7. A two-week run-in period will precede enrollment in the trial to document the indolent nature of the subjects selected; healing rate is not to be > 40% during this period.
8. Subject does not exhibit clinical signs / symptoms of infection upon gross observation or have been diagnosed with an active infection at time of screening.
9. Subject has adequate control of diabetes demonstrated by Hemoglobin A1c < 12% within 90 days of screening.
10. Subject has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days of the first screening visit:

    * Dorsal transcutaneous oxygen measurements (TCOM) ≥ 30mmHg.
    * Ankle-Brachial Index with results of ≥ 0.8 and ≤ 1.5 or had past intervention.

Exclusion Criteria:

1. Study ulcer wound surface is area greater than 25 cm2.
2. Study ulcer has > 40% wound healing during the 14 days screening period.
3. Subject has a known history of poor compliance with medical treatments.
4. Subject is presently participating in another clinical trial.
5. Subject has a known or suspected local malignancy to the Study diabetic ulcer, or systemic malignancy.
6. Subject has been diagnosed with autoimmune connective tissues diseases.
7. Subject has received graft material or topical growth factors on the study ulcer within the previous 30 days.
8. Subject has received application of topical steroids on the study ulcer surface within the previous 30 days.
9. Subject is pregnant or breast feeding.
10. Subject is on dialysis.
11. Subject is taking medications that are considered immune system modulators or cytotoxic chemotherapies.
12. Subject cannot be on systemic antibiotics prior to randomization, however, during the treatment phase infection management may include systemic antibiotics if in conjunction with debridement.
13. Subject has a known allergy to ingredients/components of AC5.
14. Subject has osteomyelitis, and/or bony prominences present in the wound.
15. Subject has ulcer probing to bone and tendon. (UT Grade II or III A-D).
16. Subject is unable to comply with planned study procedures and treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of wounds closed | before or at 12 weeks
  100% epithelialization
Change in wound area size | from randomization through to end of study (at 12 weeks) for non-closed wounds
  Assess the percent change in wound area
Days to complete wound closure | before or at 12 weeks
  median and mean

SECONDARY OUTCOMES:
Number of units used to achieve wound closure | before or at 12 weeks
  number of units used
Changes in quality of life | before or at 12 weeks
  Pain, odor, itch intensity and activities of daily living are assessed before any ulcer manipulations. Subject will fill out the quality of life form which utilizes a numeric scale from 0 (minimum) to indicate no pain, no odor, no itch, normal activities of daily living -10 (maximum) to indicate worst possible pain, extremely strong odor, worst possible itch and not able to perform activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Brock Liden, DPM, Principal Investigator — WAFL, Inc.
Locations (2):
- United States (2):
  - Dr. Christopher Gauland, Greenville, North Carolina
  - Dr. Brock Liden, Circleville, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warriner RA, Snyder RJ, Cardinal MH. Differentiating diabetic foot ulcers that are unlikely to heal by 12 weeks following achieving 50% percent area reduction at 4 weeks. Int Wound J. 2011 Dec;8(6):632-7. doi: 10.1111/j.1742-481X.2011.00860.x. Epub 2011 Sep 23. PMID 21951763
- [Background] Rahmani G, Prats J, Norchi T, Kates S, McInerney V, Woods J, Kelly J. First Safety and Performance Evaluation of T45K, a Self-Assembling Peptide Barrier Hemostatic Device, After Skin Lesion Excision. Dermatol Surg. 2018 Jul;44(7):939-948. doi: 10.1097/DSS.0000000000001468. PMID 29381543
- [Background] Koutsopoulos S. Self-assembling peptide nanofiber hydrogels in tissue engineering and regenerative medicine: Progress, design guidelines, and applications. J Biomed Mater Res A. 2016 Apr;104(4):1002-16. doi: 10.1002/jbm.a.35638. Epub 2016 Jan 25. PMID 26707893
- [Background] Kapp D, Pfendler L, D'Oro L, Wolcott R. Early clinical performance of an adaptive self-assembling barrier scaffold in nonhealing chronic wounds: a review of six cases. Wounds. 2022 Jan;33(1):20-30. doi: 10.25270/wnds/2022.2030. PMID 35108216